CLINICAL TRIAL: NCT03309956
Title: Comparison of Holter With Leadless Patch Ambulatory Electrocardiographic Monitoring in Children
Brief Title: Holter Versus Zio Patch Electrocardiographic Monitoring in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR5436
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Arrhythmias, Cardiac; Heart Block
Keywords: Ambulatory Electrocardiography; Holter Monitor; Zio Patch Monitor; Pediatrics
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Block | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: All patients will receive the same intervention, namely both devices at the same time for 48 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Holter Monitor and Zio Patch (Other): All subjects will wear the Holter monitor and Zio patch for a total of 48 hours.
  Interventions: Device: Holter Monitor; Device: Zio Patch

INTERVENTIONS:
Device: Holter Monitor — A Holter monitor is a battery-operated portable device that measures and records your heart's electrical activity (ECG) continuously. Patients in this study will wear the monitor for 48 hours.
Device: Zio Patch — The Zio Patch is a small, adhesive, water-resistant single lead electrocardiographic monitoring device. Patients in this study will wear the patch for 48 hours.

SUMMARY:
This prospective study aims to compare the diagnostic yield, or ability to detect an arrhythmia, of the traditional Holter monitor versus the novel Zio patch monitor in pediatric patients referred for ambulatory electrocardiographic (ECG) monitoring. Children will wear both devices simultaneously for 48 hours and the incidence of clinically significant arrhythmias will be compared.

DETAILED DESCRIPTION:
Patients under age 22 years at Children's Hospital of New York (CHONY) who are referred for ambulatory ECG monitoring will be consented and enrolled prospectively to have the Holter monitor and the Zio patch placed simultaneously in the pediatric cardiology clinic. Patients will be instructed to wear both devices for 48 hours. Demographic data will be collected, including date of birth, age, gender, weight, height, chest circumference, body surface area, indication for ambulatory ECG monitoring, prior congenital heart disease, prior cardiac surgery, and prior Holter or Zio patch use. A patient satisfaction survey will be given to the patient and parent/guardian after completion of the study to compare the comfort, interference with daily activities, adverse events (such as skin irritation or if either device fell off), and preference for each device. Holter monitors will be returned to the clinic along with the patient satisfaction survey, and the Zio patch will be mailed back to manufacturer headquarters and the report will be returned to the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Any patient under age 22 years who has been referred for ambulatory ECG monitoring at Children's Hospital of New York.

Exclusion Criteria:

* Any known skin allergy or sensitivity to adhesive material.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 247 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Liberman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett PM, Komatireddy R, Haaser S, Topol S, Sheard J, Encinas J, Fought AJ, Topol EJ. Comparison of 24-hour Holter monitoring with 14-day novel adhesive patch electrocardiographic monitoring. Am J Med. 2014 Jan;127(1):95.e11-7. doi: 10.1016/j.amjmed.2013.10.003. Epub 2013 Oct 15. PMID 24384108
- [Background] Bolourchi M, Batra AS. Diagnostic yield of patch ambulatory electrocardiogram monitoring in children (from a national registry). Am J Cardiol. 2015 Mar 1;115(5):630-4. doi: 10.1016/j.amjcard.2014.12.014. Epub 2014 Dec 18. PMID 25591894
- [Background] Cheung CC, Kerr CR, Krahn AD. Comparing 14-day adhesive patch with 24-h Holter monitoring. Future Cardiol. 2014 May;10(3):319-22. doi: 10.2217/fca.14.24. PMID 24976467
- [Background] Lobodzinski SS. ECG patch monitors for assessment of cardiac rhythm abnormalities. Prog Cardiovasc Dis. 2013 Sep-Oct;56(2):224-9. doi: 10.1016/j.pcad.2013.08.006. PMID 24215754
- [Background] Rosenberg MA, Samuel M, Thosani A, Zimetbaum PJ. Use of a noninvasive continuous monitoring device in the management of atrial fibrillation: a pilot study. Pacing Clin Electrophysiol. 2013 Mar;36(3):328-33. doi: 10.1111/pace.12053. Epub 2012 Dec 13. PMID 23240827
- [Background] Schreiber D, Sattar A, Drigalla D, Higgins S. Ambulatory cardiac monitoring for discharged emergency department patients with possible cardiac arrhythmias. West J Emerg Med. 2014 Mar;15(2):194-8. doi: 10.5811/westjem.2013.11.18973. PMID 24672611
- [Background] Tung CE, Su D, Turakhia MP, Lansberg MG. Diagnostic Yield of Extended Cardiac Patch Monitoring in Patients with Stroke or TIA. Front Neurol. 2015 Jan 12;5:266. doi: 10.3389/fneur.2014.00266. eCollection 2014. PMID 25628595
- [Background] Turakhia MP, Hoang DD, Zimetbaum P, Miller JD, Froelicher VF, Kumar UN, Xu X, Yang F, Heidenreich PA. Diagnostic utility of a novel leadless arrhythmia monitoring device. Am J Cardiol. 2013 Aug 15;112(4):520-4. doi: 10.1016/j.amjcard.2013.04.017. Epub 2013 May 11. PMID 23672988

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Holter Monitor and Zio Patch
Started | 247
Completed | 200
Not Completed | 47
Not completed — Devices worn for <24 hrs or >72 hrs, device failing to record, or devices were lost | 47

BASELINE CHARACTERISTICS:
Population: 247 subjects were enrolled. 47 patients were excluded from the arrhythmia analysis due to one or both devices being worn for <24 hours (n = 18) or >72 hours (n = 4), either device failing to record (n = 11), or one or both devices being lost (n = 14). A total of 200 patients completed the study and were included for the arrhythmia analysis after attrition. The Baseline Population characteristics are reported for the final 200 participants.
Groups:
- Holter Monitor and Zio Patch: All subjects will wear the Holter monitor and Zio patch for a total of 48 hours.
  Holter Monitor: A Holter monitor is a battery-operated portable device that measures and records your heart's electrical activity (ECG) continuously. Patients in this study will wear the monitor for 48 hours.
  Zio Patch: The Zio Patch is a small, adhesive, water-resistant single lead electrocardiographic monitoring device. Patients in this study will wear the patch for 48 hours.
  247 subjects were enrolled. 47 patients were excluded from the arrhythmia analysis due to one or both devices being worn for <24 hours (n = 18) or >72 hours (n = 4), either device failing to record (n = 11), or one or both devices being lost (n = 14). A total of 200 patients completed the study and were included for the arrhythmia analysis after attrition. The Baseline Population characteristics are reported for the final 200 participants.
Arm/Group | Holter Monitor and Zio Patch
Number analyzed (Participants) | 200
Age, Customized [Count of Participants; unit: Participants]
  0-7 years old | 40
  8-17 years old | 160
  18-65 years old | 0
  >65 years old | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 200
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 200
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Difference in Detection of Clinically Significant Arrhythmias for the Zio Versus the Holter
Description: The diagnostic yield, or the ability to detect an arrhythmia, will be measured for the Holter monitor and the Zio patch monitor for each patient. The diagnostic yield for each arrhythmia subtype will be determined for each device across all patients and compared in paired statistical analysis (McNemar's test).
Time Frame: 48 hours
Population: 247 subjects were enrolled. 47 patients were excluded from the arrhythmia analysis due to one or both devices being worn for <24 hours (n = 18) or >72 hours (n = 4), either device failing to record (n = 11), or one or both devices being lost (n = 14). A total of 200 patients completed the study and were included for the arrhythmia analysis after attrition.
Measure: Number; unit: participants
Arm/Group | Holter Monitor and Zio Patch
Number analyzed (Participants) | 200
participants | 0
Statistical Analysis 1: Comparison: Holter Monitor and Zio Patch; Test type: Superiority; p = 0.23, McNemar

2. Secondary Outcome: Prevalence of Artifact Detected
Description: The aggregate percent analyzable data of the Holter monitor compared to the Zio Patch across all patients will be calculated using descriptive statistics.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of artifact detected
Groups:
- Holter Monitor: All subjects will wear the Holter monitor and Zio patch for a total of 48 hours.
  Holter Monitor: A Holter monitor is a battery-operated portable device that measures and records your heart's electrical activity (ECG) continuously. Patients in this study will wear the monitor for 48 hours.
- Zio Patch: All subjects will wear the Holter monitor and Zio patch for a total of 48 hours.
  Zio Patch: The Zio Patch is a small, adhesive, water-resistant single lead electrocardiographic monitoring device. Patients in this study will wear the patch for 48 hours.
Arm/Group | Holter Monitor | Zio Patch
Number analyzed (Participants) | 200 | 200
percentage of artifact detected | 5.6 [2.4 to 15.7] | 2.8 [1.1 to 8.6]

3. Other Pre Specified Outcome: Percentage of Patients Who Preferred the Zio Over the Holter
Description: Descriptive statistics will be used to analyze survey results. A one page patient satisfaction survey will be filled out at the end of the 48 hours to compare patient/parental preference and possible adverse reactions for each device.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Monitor and Zio Patch
Number analyzed (Participants) | 200
Participants | 150

ADVERSE EVENTS:
Time Frame: Up to 48 hours
Description: 247 subjects were enrolled. 47 patients were excluded from the arrhythmia analysis due to one or both devices being worn for <24 hours (n = 18) or >72 hours (n = 4), either device failing to record (n = 11), or one or both devices being lost (n = 14). A total of 200 patients completed the study and were included for the arrhythmia analysis after attrition. Adverse Events were monitored and reported for the final 200 participants.
Arm/Group | Holter Monitor and Zio Patch
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT03309956/Prot_SAP_000.pdf